CLINICAL TRIAL: NCT06986434
Title: A Clinical Study on the Safety and Efficacy of CAR19-BCMA Dual-target CAR-T Cell Therapy for Relapsed/Refractory Plasma Cell Neoplasms
Brief Title: CAR19BCMA CAR-T Cells for the Treatment of R/R Plasma Cell Neoplasms
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR19BCMA-XYBYXB
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Plasma Cell Neoplasms
Keywords: CAR-T; plasma cell neoplasms; CD19/BCMA
MeSH Terms: conditions — Recurrence; Neoplasms, Plasma Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This is a single arm treatment of CAR19BCMA CAR-T cell (Experimental): Experimental: CAR19BCMA-T cells Therapy Investigational product: CAR19BCMA-T cells Route of administration: Intravenous injection Lymphodepleting chemotherapy regimen: A combination of fludarabine and cyclophosphamide will be administered prior to the infusion of CD19BCMA-CAR-T cells.
  Interventions: Genetic: CAR19BCMA-T cells; Drug: fludarabine and cyclophosphamide

INTERVENTIONS:
Genetic: CAR19BCMA-T cells — CAR19BCMA-T cells Each subject will be infused with single dose of CD19BCMA-CAR-T cells. A classic "3+3" dose escalation will be employed. The low dose is 1×10^6 /kg, the medium dose is 2×10^6 /kg, and the high dose is 3×10^6 /kg.
Drug: fludarabine and cyclophosphamide — Drug: Fludarabine Fludarabine will be given at a dose of 30 mg/m2/day intravenously (IV) for 3 days prior to the infusion of CD19BCMA-CAR-T cells.
  Drug: Cyclophosphamide Cyclophosphamide will be given at a dose of 300 mg/m2/day intravenously (IV) for 3 days prior to the infusion of CD19BCMA-CAR-T cells.

SUMMARY:
This is a single arm study to evaluate the safety and efficacy of CAR19BCMA CAR-T cells in the treatment of relapsed/refractory CD19/BCMA positive plasma cell neoplasms.

DETAILED DESCRIPTION:
This study is an exploratory clinical trial of a single-arm, open, single-center treatment of CAR19BCMA CAR-T cell. 20 subjects with relapsed or refractory CD19/ BCMA positive positive plasma cell neoplasms will be enrolled and received CAR19BCMA CAR T cells injection therapy, and related data such as adverse reactions and therapeutic effects after medication were followed up. To evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

Relapsed/refractory CD19BCMA positive plasma cell neoplasms must be assured and meet all of the following conditions:

①Confirmation for either BCMA or CD19 positivity using immunohistochemistry or flow cytometry.

②Patients with multiple myeloma, plasma cell carcinoma, and plasma cell leukemia who have received at least three 3 lines treatment (including anti-CD38 monoclonal antibodies, protease inhibitors, immunosuppressants, etc.) but have failed or experienced relapse.

③Patients with system light chain amyloidosis who have received at least 2 lines treatments in the past [anti-CD38 monoclonal antibody, proteasome inhibitor (PI), or immunomodulatory drug (IMiD)], but have failed or experienced relapse.

Age 18-80 years, no gender restrictions; ECOG score ≤ 2 points; Expected survival period is not less than 3 months; HGB≥60g/L; Liver function and cardiopulmonary function meet the following requirements: (1) left ventricular ejection fraction≥50%; (2) Oxygen saturation >90%; (3)Total bilirubin ≤1.5×ULN, ALT and AST≤2.5×ULN; Participants agreed to use contraception from the time of informed consent until 1 year after CAR-T cell infusion.

Exclusion Criteria:

Severe heart failure with left ventricular ejection fraction <50%; A history of severe lung function impairment; Combined with other advanced malignant tumors; Complicated with severe infection that could not be effectively controlled; Severe autoimmune disease or congenital immune deficiency; Active hepatitis (hepatitis B virus DNA [HBV-DNA] or hepatitis C virus RNA [HCV-RNA] test results above the lower limit of detection); Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection; History of severe allergy to biological products (including antibiotics); Patients with other serious physical or mental illnesses or laboratory abnormalities that could increase the risk of participating in the study or interfere with the results of the study, and those who were deemed by the investigator to be unsuitable for participation in the study.

Female patients (those with fertility) are in pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-26 (Estimated); Primary Completion 2027-05-22 (Estimated); Study Completion 2028-08-25 (Estimated)

PRIMARY OUTCOMES:
According to the incidence of treatment-related adverse events (AEs) to evaluate the safetyof CAR19BCMA CAR-T cells in the treatment of relapsed/refractory CD19+BCMA+plasma cell neoplasms. | up to 3 years
  Incidence of treatment-related adverse events (AEs) Description: Number and severity of adverse events graded according to CTCAE v5.0, including cytokine release syndrome (CRS) graded by ASTCT criteria and immune effector cell-associated neurotoxicity syndrome (ICANS) graded by ASBMT criteria
According to the determine the Maximal Tolerable Dose(MTD) to evaluate the safety of CAR19BCMA CAR-T cells in the treatment of relapsed/refractory CD19+BCMA+ plasma cell neoplasms. | MTD will be determined based on DLTs observed during the first 28 days of study treatment

SECONDARY OUTCOMES:
According to the objective response rate (ORR) to evaluate the efficacy of CAR19BCMA CAR-T cells in the treatment of relapsed/refractory CD19+BCMA+ plasma cell neoplasms. | Within 3 months following infusion of CAR19BCMA CAR-T cells
  Overall response rate (ORR) Description: Multiple myeloma (plasma cell neoplasms, plasma cell leukemia) refers to the efficacy evaluation criteria in the Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma (revised in 2024),ORR includes strictly defined proportions of complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), and minimal response (MR).

OTHER OUTCOMES:
According to the pharmacokinetics (number of CAR-T cells in peripheral blood was measured to evaluate the persistence of CAR-T cells) to explore the kinetics and clonal evolution of CAR19BCMA CAR-T cells. | Up to 12 months after CAR-T treatment

CONTACTS AND LOCATIONS:
Locations (1):
- the Fifth Medical Center of Chinese People's Liberation Army General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No